CLINICAL TRIAL: NCT01622361
Title: A Phase III, Open-Label, Prospective, Randomized, Multicenter, Neo-adjuvant Study of Chemotherapy Versus Endocrine Therapy in Premenopausal Patient With Hormone Responsive, HER2 Negative, Lymph Node Positive Breast Cancer
Brief Title: Premenopausal Patient With Hormone Responsive, HER2 Negative, Lymph Node Positive Breast Cancer
Acronym: NEST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Breast Cancer Study Group (Other)
Responsible Party: Principal Investigator, Sei-Hyun Ahn, M.D., Ph.D., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG012
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant; endocrine therapy; premenopausal; hormone responsive; HER2 negative; lymph node positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy Group (Active Comparator): Chemotherapy Adriamycin+Cyclophosphamide>Docetaxel
  Interventions: Drug: Adriamycin+Cyclophosphamide>Docetaxel
- Endocrine therapy group (Experimental): Endocrine therapy(GnRHa with Tamoxifen) group
  Interventions: Drug: GnRHa with Tamoxifen

INTERVENTIONS:
Drug: Adriamycin+Cyclophosphamide>Docetaxel — 1. Adriamycin 60mg/m2 + Cyclophosphamide 600mg/m2
     * Route: by slow intravenous bolus
     * Schedule: every 3weeks for 4 cycle
  2. Docetaxel 75mg/m2
     * Route: intravenous as per local practice
     * Schedule: every 3weeks for 4 cycle
  Other Names: Chemotherapy
  Arms: Chemotherapy Group
Drug: GnRHa with Tamoxifen — 1. Goserelin(GnRHa) 3.6mg
     * Route: subcutaneously under the abdominal skin
     * Schedule: every 4weeks for 6cycles (period of 34 days between 2 administrations must not be exceeded)
  2. Tamoxifen 20mg/day
     * Route: Oral
     * Schedule: everyday
  Other Names: Endocrine Therapy
  Arms: Endocrine therapy group

SUMMARY:
The purpose of this study is to compare neo-adjuvant therapy of cytotoxic chemotherapy versus GnRHa with tamoxifen , of response rate(RR) in patients of hormone responsive and HER2 negative, lymph node positive, primary breast cancer in premenopausal women.

DETAILED DESCRIPTION:
1. Primary objective

   : Response Rate-MRI and/or Caliper
2. Secondary objectives

   * Pathologic complete response
   * Rate of conservation surgery
   * Ki-67 changes and its relationship to treatment response
   * Length of time to maximum response within the treatment period
   * Tolerability of two treatments
   * Disease-free survival(DFS)
   * Overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary invasive breast cancer which is thought to be suitable for neo-adjuvant treatment
2. Pathologically proven lymph node positive tumor(FNAB or Core biopsy)
3. Tumor must be ER positive(eligible patients include Allred score 5 and more, Modified Allred 4 and more) and HER-2 negative(IHC score is 0-1+; If IHC score is 2+, the result of FISH or SISH is negative)
4. Premenopausal women

   Premenopausal status as defined by :
   * Last menses within 6 month of randomization or
   * For patients who have had a unilateral oophorectomy, E2 ≥ 20PG/mL and FSH < 30mIU/Ml within 4 weeks of randomization
5. over 20 years old
6. Pre-treatment haematology and biochemistry values within acceptable limits :

   * ANC ≥ 1.5 × 109/l
   * Hb > 9g/dl
   * Platelets ≥ 100 × 109/l
   * AST/ALT ≤ 1.5 × ULN(Upper Limit of Normal)
   * ALP ≤ 1.5 × ULN
   * Serum bilirubin ≤ 1.5 × ULN
   * Serum creatinine ≤ 1.5 × ULN
7. ECOG PS of 0 or 1
8. No concomitant medical, psychiatric or geographic problems that might prevent completion of treatment or follow-up
9. Before any study-specific procedures, the appropriate written informed consent must be obtained

Exclusion Criteria:

1. Inflammatory breast cancer
2. Inoperable disease that is judged very unlikely to be rendered operable by neo-adjuvant treatment
3. Known severe hypersensitivity to GnRHa treatment
4. Bilateral invasive breast cancer
5. Other serious illness or medical condition:

   * congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrhythmias
   * history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
   * active uncontrolled infection
6. HRT within 4 weeks of starting treatment
7. Definite contra-indications for the use of corticosteroids.
8. Last 10 years with a history of other malignant tumor (except in the case of basal cell carcinoma or cervical carcinoma in situ, and where treatment consisted solely of resection)
9. Systemic metastatic (Tests for the diagnosis of systemic metastatic comply with the guideline in each institution)
10. Pregnant or breastfeeding women
11. Chronic oral treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 20 mg methylprednisolone or equivalent).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6 months

SECONDARY OUTCOMES:
Pathologic complete response | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Gwark S, Noh WC, Ahn SH, Lee ES, Jung Y, Kim LS, Han W, Nam SJ, Gong G, Kim SO, Kim HJ. Axillary Lymph Node Dissection Rates and Prognosis From Phase III Neoadjuvant Systemic Trial Comparing Neoadjuvant Chemotherapy With Neoadjuvant Endocrine Therapy in Pre-Menopausal Patients With Estrogen Receptor-Positive and HER2-Negative, Lymph Node-Positive Breast Cancer. Front Oncol. 2021 Sep 30;11:741120. doi: 10.3389/fonc.2021.741120. eCollection 2021. PMID 34660302
- [Derived] Gwark S, Ahn SH, Noh WC, Lee ES, Jung Y, Kim LS, Han W, Nam SJ, Gong G, Kim SO, Kim HJ. Patient-Reported Outcomes From Phase III Neoadjuvant Systemic Trial Comparing Neoadjuvant Chemotherapy With Neoadjuvant Endocrine Therapy in Pre-Menopausal Patients With Estrogen Receptor-Positive and HER2-Negative, Lymph Node-Positive Breast Cancer. Front Oncol. 2021 Jul 2;11:608207. doi: 10.3389/fonc.2021.608207. eCollection 2021. PMID 34277393
- [Derived] Kim HJ, Noh WC, Lee ES, Jung YS, Kim LS, Han W, Nam SJ, Gong G-, Kim HJ, Ahn SH. Efficacy of neoadjuvant endocrine therapy compared with neoadjuvant chemotherapy in pre-menopausal patients with oestrogen receptor-positive and HER2-negative, lymph node-positive breast cancer. Breast Cancer Res. 2020 May 27;22(1):54. doi: 10.1186/s13058-020-01288-5. PMID 32460816